CLINICAL TRIAL: NCT00528697
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Dose-Ranging Study of the Safety and Efficacy of ABT-089 in Children With Attention Deficit-Hyperactivity Disorder (ADHD)
Brief Title: A Safety and Efficacy Study of ABT-089 in Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-888
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — pozanicline; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): Lowest ABT-089 dose
  Interventions: Drug: ABT-089
- 2 (Experimental): Low-medium ABT-089 dose
  Interventions: Drug: ABT-089
- 3 (Experimental): Medium-high ABT-089 dose
  Interventions: Drug: ABT-089
- 4 (Experimental): Highest ABT-089 dose
  Interventions: Drug: ABT-089
- 5 (Active Comparator): atomoxetine
  Interventions: Drug: atomoxetine
- 6 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ABT-089 — Subjects will take 0.5 and 1 and/or 5 and/or 10 mg ABT-089 tablets (actual dose based on weight) once daily for 8 weeks.
  Arms: 1; 2; 3; 4
Drug: atomoxetine — Subjects will take 10, and/or 18 and/or 25 mg atomoxetine tablets once daily for 8 weeks.
  Arms: 5
Drug: placebo — Subject will take a tablet once daily for 8 weeks
  Arms: 6

SUMMARY:
The purpose of this study is to test if the investigational medication ABT-089 is a safe and effective treatment for children with Attention-Deficit/Hyperactivity Disorder or ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily signed an informed consent form
* Meet diagnostic criteria for attention-deficit/hyperactivity disorder (ADHD) based on detailed evaluation and interview with parent(s)
* First grade or higher in a school setting 3 days/week
* Subject is generally in good health based on medical history, physical examination, clinical lab tests, and ECG
* Subject weighs at least 37 pounds (17 kg)
* Female subjects of childbearing potential must have a negative urine pregnancy test at screening and baseline and agree to comply with applicable contraceptive requirements
* Subject and parents have been judged by the study doctor to be reliable to keep required appointments for clinic visits and all tests, including blood draws, and examinations

Exclusion Criteria:

* Subject is not functioning at an age-appropriate level intellectually
* Subject has a current or past diagnosis of bipolar disorder, psychosis, autism, Asperger's syndrome, or pervasive developmental disorder
* Current diagnosis of obsessive-compulsive disorder, eating disorder, anxiety disorder or depressive disorder requiring treatment of any kind
* Subject has a history of significant allergic reaction to any drug
* Subject requires ongoing treatment with any psychiatric medication
* Subject has a serious medical condition, seizure disorder (except febrile seizures as an infant), or history of substance abuse or dependence

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
ADHD-RS-IV (HV) - Administered by study doctor | Screening, Day -1, Day 7, Day 14, Day 28, Day 42, Day 56

SECONDARY OUTCOMES:
Health Outcomes Measurements | Baseline to Final Evaluation of 8-week treatment period
Clinical Global Impression-ADHD-Severity Scale | Baseline to Final Evaluation of 8-week treatment period
Parent Rating Scales | Baseline to Final Evaluation of 8-week treatment period
Teacher Rating Scale | Baseline to Final Evaluation of 8-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gault, MD, PhD, MD, Study Director — AbbVie
Locations (20):
- United States (20):
  - Site Reference ID/Investigator# 5999, Little Rock, Arkansas
  - Site Reference ID/Investigator# 5979, El Centro, California
  - Site Reference ID/Investigator# 5986, Boulder, Colorado
  - Site Reference ID/Investigator# 5993, Bradenton, Florida
  - Site Reference ID/Investigator# 5995, Jacksonville, Florida
  - Site Reference ID/Investigator# 5977, Orlando, Florida
  - Site Reference ID/Investigator# 5981, Northbrook, Illinois
  - Site Reference ID/Investigator# 5982, Overland Park, Kansas
  - Site Reference ID/Investigator# 5992, Omaha, Nebraska
  - Site Reference ID/Investigator# 5997, Las Vegas, Nevada
  - Site Reference ID/Investigator# 5987, Clementon, New Jersey
  - Site Reference ID/Investigator# 5996, Eugene, Oregon
  - Site Reference ID/Investigator# 5984, Portland, Oregon
  - Site Reference ID/Investigator# 5980, Salem, Oregon
  - Site Reference ID/Investigator# 5994, Charleston, South Carolina
  - Site Reference ID/Investigator# 5976, Memphis, Tennessee
  - Site Reference ID/Investigator# 6000, Austin, Texas
  - Site Reference ID/Investigator# 5998, Herndon, Virginia
  - Site Reference ID/Investigator# 5978, Bellevue, Washington
  - Site Reference ID/Investigator# 5983, Middleton, Wisconsin

REFERENCES:
- [Derived] Wilens TE, Gault LM, Childress A, Kratochvil CJ, Bensman L, Hall CM, Olson E, Robieson WZ, Garimella TS, Abi-Saab WM, Apostol G, Saltarelli MD. Safety and efficacy of ABT-089 in pediatric attention-deficit/hyperactivity disorder: results from two randomized placebo-controlled clinical trials. J Am Acad Child Adolesc Psychiatry. 2011 Jan;50(1):73-84.e1. doi: 10.1016/j.jaac.2010.10.001. Epub 2010 Nov 25. PMID 21156272